CLINICAL TRIAL: NCT04954599
Title: Phase 1/2 Modular Dose Escalation With Cohort Expansion of CP-506 (HAP) in Patients With Solid Tumor Types With High Incidence of HRD/FAD in Monotherapy or With Carboplatin or Patients With Solid Tumour and OPD Receiving ICI
Brief Title: Phase 1/2 Clinical Trial of CP-506 (HAP) in Monotherapy or With Carboplatin or ICI
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other); Jules Bordet Institute (Other); Academisch Ziekenhuis Maastricht (Other); Vall d'Hebron Institute of Oncology (Other); University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TUMAGNOSTIC(CP506-001); 2021-000423-12 (EudraCT Number); 694812 (Other Grant/Funding Number: Horizon 2020 Framework Programme)
Record Dates: First submitted 2021-06-16; First posted 2021-07-08 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: Homologous recombination DNA repair defects; Fanconi Anaemia DNA repair defects; Triple negative breast cancer; Ovarian cancer; Prostate cancer; Pancreatic cancer; Head and neck cancer; Hypoxia Activated Prodrug; Alkylating Agents; Carboplatin; Immune Checkpoint Inhibitor
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Pancreatic Neoplasms; Head and Neck Neoplasms | interventions — Carboplatin; Immune Checkpoint Inhibitors; Ipilimumab; Nivolumab; pembrolizumab; atezolizumab; avelumab; durvalumab; cemiplimab

STUDY DESIGN:
Intervention Model Description: A modular, multi-arm, multi-part, first time in patient study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Module 1A Monotherapy Multiple Ascending Dose (Experimental): Multiple ascending dose cohorts dosing CP-506 monotherapy in all patients up to a maximally tolerated or maximally feasible dose Intervention: Drug: CP-506
  Interventions: Drug: CP-506
- Module 1B Monotherapy Dose Expansion Cohort (Experimental): Expansion cohort dosing CP-506 monotherapy in patients at recommended phase 2 dose (RP2D) Intervention: Drug: CP-506
  Interventions: Drug: CP-506
- Module 2A Combination with carboplatin Multiple Ascending Dose (Experimental): Multiple ascending dose cohorts dosing CP-506 in combination with carboplatin in all patients up to a maximally tolerated or maximally feasible dose Intervention: Drug: CP-506
  Interventions: Drug: CP-506; Drug: Carboplatin
- Module 2B Combination with carboplatin Dose Expansion Cohort (Experimental): Expansion cohort dosing CP-506 in combination with carboplatin in patients at recommended phase 2 dose (RP2D) Intervention: Drug: CP-506
  Interventions: Drug: CP-506; Drug: Carboplatin
- Module 3A Combination with Immune Checkpoint Inhibitor Multiple Ascending Dose (Experimental): Multiple ascending dose cohorts dosing CP-506 in combination with Immune Checkpoint Inhibitor in all patients up to a maximally tolerated or maximally feasible dose Intervention: Drug: CP-506
  Interventions: Drug: CP-506; Drug: Immune checkpoint inhibitor
- Module 3B Combination with carboplatin Dose Expansion Cohort (Experimental): Expansion cohort dosing CP-506 in combination with Immune Checkpoint Inhibitor in patients at recommended phase 2 dose (RP2D) Intervention: Drug: CP-506
  Interventions: Drug: CP-506; Drug: Immune checkpoint inhibitor

INTERVENTIONS:
Drug: CP-506 — CP-506 is a hypoxia-activated DNA alkylating agent specifically designed to have a bystander effect, aqueous solubility, oral bioavailability, and no off-mechanism activation by the human aerobic reductase AKR1C3
  Other Names: HAP CP-506
Drug: Carboplatin — Antineoplastic agent, ATC Code: LO1X A02
  Other Names: Paraplatin
  Arms: Module 2A Combination with carboplatin Multiple Ascending Dose; Module 2B Combination with carboplatin Dose Expansion Cohort
Drug: Immune checkpoint inhibitor — Drug that blocks immune checkpoint proteins: PD-1, PD-L1, CTLA-4
  Other Names: Ipilimumab; Nivolumab; Pembrolizumab; Atezolizumab; Avelumab; Durvalumab; Cemiplimab
  Arms: Module 3A Combination with Immune Checkpoint Inhibitor Multiple Ascending Dose; Module 3B Combination with carboplatin Dose Expansion Cohort

SUMMARY:
A modular, first time in human, open label, multiple dose, accelerated escalation with cohort expansion study of the safety and pharmacokinetics of intravenous infusion of CP-506, a tumor agnostic Hypoxia Activated Prodrug in patients with HRD/FAD solid tumours or tumor types with high incidence of HRD/FAD in monotherapy or in combination with carboplatin or patients with solid tumour and oligoprogressive disease receiving immune checkpoint inhibitors (ICI): a phase I-IIa clinical trial

DETAILED DESCRIPTION:
This study is a First in Human, early phase (I/IIa), 3 modules, 2 parts (A- dose escalation and B- cohort expansion), open-label, uncontrolled, multi-center, multiple dose, accelerated 3+3 dose escalation study. The study consist of 3 study modules. Module 1 is monotherapy with accelerated dose escalation. Modules 2 and 3 are also accelerated dose escalation modules, but with a combination of CP-506 with either Carboplatin or ICI. Initiation of modules 2 and 3 are dependent on the decision by the Independent Data Monitoring Committee (IDMC) based on the safety, tolerability and feasibility information from the study as a whole.

Each study modules will consist of a Part A (dose finding) and an optional Part B (cohort expansion). The option to start Part B will be decided by the IDMC based on safety, tolerability and feasibility information from the study as a whole. The expansion cohorts will explore preliminary efficacy.

Modules 2 and 3 will start after completion of module 1 and definition of the "minimal biological effective dose" (MBED) as the dose that results in 1) a decrease of 20% of hypoxia radiomics score on sequential CT of at least one lesion OR 2) a decrease of 20% of the initial tumour volume of at least one lesion.

MBED is assessed by CT scan at visit 7, 12 and 13. After observation of an MBED in three patients, the data supporting the MBED assessment will be reviewed by the IDMC for confirmation.

A maximum of 126 patients with advanced or metastatic cancer will be recruited in this study.

* Module 1 - Monotherapy: up to 24 patients for Part A and 10 patients for Part B for whom no standard of care or known effective treatment options are available and with cancers that show a considerable incidence of Homologous Recombination or Fanconi Anaemia DNA repair defects (HRD/FAD)
* Module 2 - Combination with Carboplatin: up to 24 patients for Part A and 22 patients for Part B for patients that receive carboplatin as standard of care: triple negative breast cancer and ovarian cancer.
* Module 3 - Combination with ICI: up to 24 patients for Part A and 22 patients for Part B with advanced or metastatic cancer for whom standard of care immune checkpoint inhibitor (ICI) are currently administered for at least 6 months, would still be administered according to the treating clinician, outside any clinical trial but resulted in oligoprogression.

The complete CP-506 therapy consists of three cycles of CP-506 treatment. Each treatment cycle consists of three consecutive days of IV infusion for two hours and one day for observation and blood sampling, and a recovery time of 3 weeks. Patients are expected to come to the hospital for 18 visits. They consist of 1 screening visit, 3 cycles of CP-506 treatment. Each cycle will be followed by a post cycle visit after 14 and 21 days. The follow up visit will take place at day 105.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 years or more at the time of signing the informed consent
2. Be willing and able to provide written informed consent for the trial
3. Life expectancy of at least 3 months
4. Be willing to have a biopsy collection procedure
5. ECOG Performance status <= 2
6. Must have adequate organ and bone marrow function, defined as the following:

   6.1. ANC ≥ 1500 µL 6.2. Hemoglobin ≥ 9.0 g/dL 6.3. Platelets ≥ 100 000 µL 6.4. Total bilirubin ≤ 1.5 × ULN OR direct bilirubin ≤ ULN for participants with total bilirubin levels >1.5 × ULN 6.5. AST (SGOT) and ALT (SGPT) ≤ 2.5 × ULN (≤ 5 × ULN for participants with liver metastases) 6.6. Creatinine ≤ 1.5 × ULN 6.7. Coagulation: INR ≤ 1.5 × ULN (or within therapeutic ranges for participants on anticoagulant treatment)
7. Measurable disease on CT scan (RECIST 1.1)
8. If female, not pregnant, not breastfeeding, and at least one of the following conditions applies:

   8.1. Not a woman of childbearing potential (WOCBP) 8.2. A WOCBP who agrees to follow contraceptive guidance during the treatment period and for at least 4 weeks after the last dose of study treatment and shows a negative pregnancy test before the start of the treatment
9. If male, must agree to use contraception during the treatment period and for at least 4 weeks after the last dose of study treatment
10. Able and willing to comply with the protocol Module 1 - monotherapy
11. Have histologically or cytologically-confirmed advanced or metastatic solid tumour for whom no standard of care or known effective treatment options are available
12. Have indications of Homologous Recombination (HR) or Fanconi Anaemia (FA) DNA damage repair defects, based on hereditary cancer diagnostics (e.g. BRCA1/2 carriers), dedicated HRD genomic assays (including exome-sequencing) from liquid or tissue biopsies. Presence of such a defect must have been established via a tissue based next generation sequencing test, performed --in a CAP/CLIAcertified (or comparable local or regional certification) laboratory, or via a germline test from one of the following approved providers: Myriad Genetics; Invitae; Ambry; Quest; Color Genomics; MSKCC-IMPACT; GeneDx; Foundation Medicine OR Have cancers with an increased incidence of HRD/FAD: ovarian (41%), breast (18%), pancreas (10%), prostate (9%), and head and neck (5%) OR Patients who were previously responsive to alkylating agent (Partial Response/Complete Response according to RECIST criteria).

    Module 2 - Carboplatin combination
13. Patient must be eligible to carboplatin treatment.
14. Have histologically or cytologically-confirmed advanced or metastatic solid tumour for whom no standard of care or known effective treatment options are available.
15. Receive carboplatin as standard of care: triple negative breast cancer or ovarian cancer.

    Module 3 - ICI combination
16. Have histologically or cytologically-confirmed advanced or metastatic solid tumour
17. Receiving immune checkpoint inhibitor (ICI) monotherapy as standard of care for at least 6 months prior to the beginning of the study and who are oligoprogressive. Oligoprogression disease is defined as localized treatment failure at one or two anatomic sites, with one to five progressive and measurable (according to RECIST 1.1) lesions, either new or with ≥ 20% growth of their longest diameter (short-axis in lymph nodes), while other tumor manifestations could shrink or grow less than 20% in diameter

Exclusion Criteria:

Core:

1. Prior radiotherapy to more than 25% of bone marrow
2. Not recovered from all acute toxic effects of prior anticancer therapy (excluding CTCAE Grade 1 alopecia or peripheral neuropathy)
3. Patients with significant cardiac co-morbidity, such as NYHA Class III or IV CHF, unstable angina, MI within the previous 6 months, or ventricular arrhythmias requiring drug therapy, pacemaker or implanted defibrillator. Serious, uncontrolled cardiac arrhythmia or clinically significant electrocardiogram abnormalities including second degree (Type II) or third-degree atrioventricular block. This does not apply to patient with a pace maker. Cardiomyopathy, myocardial infarction, acute coronary syndromes (including unstable angina pectoris), coronary angioplasty, stenting or bypass grafting. Congestive heart failure (Class II, III, or IV) as defined by the New York Heart Association functional classification system. Symptomatic pericarditis
4. A marked baseline prolongation of QT/QTc interval (> 450 ms)
5. History of risk factors for Torsade de Pointe (e.g. heart failure, hypokalemia, family history of Long QT syndrome)
6. Use of concomitant medication prolonging the QT/QTc interval
7. Evidence of uncontrolled infection or infection requiring a concomitant parenteral antibiotic
8. Evidence of any other significant clinical disorder or laboratory finding that in the opinion of the Investigator may compromise patient safety during study participation.
9. Patients with a diagnosis (or strong suspicion) of a rare genetic disorder related to germline biallelic HR/FA and DNA repair gene mutations, such as Fanconi anemia patients of any subtype, Ataxia telangiectasia, Xeroderma pigmentosum, Cockayne, Nijmegen breakage, Werner and Bloom syndrome patients
10. Patient or physician plans concomitant chemotherapy, radiation therapy, hormonal and/or biological treatment for cancer including immunotherapy while on study
11. Patient has been treated with any investigational drug or investigational therapeutic device within 30 days (60 days in case of biological compound) of initiating study treatment
12. Less than 4 weeks since prior major surgery
13. Known positive for HIV, Hepatitis B surface antigen positive or Hepatitis C positive with abnormal liver function tests
14. Known allergy to alkylating agents
15. Central nervous system (CNS) metastases, with the following exception:
16. Participants with asymptomatic CNS metastases who are clinically stable and have no requirement for steroids for at least 14 days prior to randomization. Note: Participants with carcinomatous meningitis or leptomeningeal spread are excluded regardless of clinical stability
17. Invasive malignancy or history of invasive malignancy other than disease under study within the last 3 years, except as noted below:

    17.1. Any other invasive malignancy for which the participant was definitively treated, has been disease-free for ≤ 3 years and in the opinion of the principal investigator will not affect the evaluation of the effects of the study treatment on the currently targeted malignancy, may be included in this clinical study 17.2. Curatively treated non-melanoma skin cancer or successfully treated in situ carcinoma 17.3. Low-risk early-stage prostate cancer defined as follows: Stage T1c or T2a with a Gleason score ≤ 6 and prostatic-specific antigen <10 ng/mL either treated with definitive intent or untreated in active surveillance that has been stable for the past year prior to randomization
18. Autoimmune disease (current or history; refer to Table 19) or syndrome that required systemic treatment within the past 2 years Note: Replacement therapies which include physiological doses of corticosteroids for treatment of endocrinopathies (for example, adrenal insufficiency) are not considered systemic treatments
19. Has a diagnosis of immunodeficiency or is receiving systemic steroids (>10 mg oral prednisone per day or equivalent) or other immunosuppressive agents within 7 days prior to randomization Note:

    19.1. Physiologic doses of corticosteroids for treatment of endocrinopathies or steroids with minimal systemic absorption, including topical, inhaled, or intranasal corticosteroids may be continued if the participant is on a stable dose, up to a maximum of 10 mg prednisone per day or equivalent 19.2. Steroids as premedication for hypersensitivity reactions (e.g., computed tomography [CT] scan premedication) are permitted.
20. Receipt of any live vaccine within 30 days prior randomization
21. Prior allogeneic/autologous bone marrow or solid organ transplantation
22. Has current pneumonitis or history of non-infectious pneumonitis that required steroids or other immunosuppressive agents Note: post-radiation changes in the lung related to prior radiotherapy and/or asymptomatic radiation-induced pneumonitis not requiring treatment (Grade 1) may be permitted if agreed upon by the investigator and Medical Monitor.
23. Recent history (within the past 6 months) of uncontrolled symptomatic ascites, pleural or pericardial effusions
24. Recent history (within the past 6 months) of gastrointestinal obstruction that required surgery, acute diverticulitis, inflammatory bowel disease, or intraabdominal abscess
25. Recent history of allergen desensitization therapy within 4 weeks of randomization
26. Cirrhosis or current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice. Note: Stable non-cirrhotic, chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) or hepatobiliary involvement of malignancy is acceptable if participant otherwise meets entry criteria
27. Known history of active tuberculosis
28. Any psychiatric disorder, or other condition that could interfere with participant's safety, obtaining informed consent, or compliance to the study procedures in the opinion of the investigator Module 1 - monotherapy
29. Patients who have received anticancer therapy (including radiotherapy) within 4 weeks of inclusion Module 2 - Carboplatin combination
30. Patients who have received anticancer therapy (including radiotherapy) within 4 weeks of inclusion with exclusion of carboplatin.

    Module 3 - ICI combination
31. Patients who have received anticancer therapy (including radiotherapy) within 4 weeks of inclusion with exception of ICI
32. Patients progressive under ICI justifying the immediate discontinuation of ICI
33. Patients who would not receive further treatment with ICI as standard of care
34. Patients with Complete Response under ICI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events including dose-limiting toxicities | Baseline until 60 days after last administration of CP-506
  The proportion of patients with treatment-emergent (serious) adverse events including dose-limiting toxicity (DLT)
Incidence of clinically significant abnormal measurements in physical examination, vital signs, electrocardiogram (ECG), lab tests and ECOG performance status | Baseline until 60 days after last administration of CP-506
  Physical examination; vital signs; electrocardiogram (ECG); haematology; clinical chemistry; urinalysis; plasma/renal makers; tumour markers; ECOG performance status

SECONDARY OUTCOMES:
Area under curve of CP-506 plasma concentration | At the end of cycle 1 day 4
  Measurement of CP-506 levels in plasma over time to calculate AUC Area under the curve (AUC) of CP-506 plasma concentration
Determine the minimal biological effective dose | Baseline until 60 days after last administration of CP-506
  Number of patients that show 1) a decrease of 20% of hypoxia radiomics score on sequential CT of at least one lesion OR 2) a decrease of 20% of the initial tumour volume of at least one lesion
Objective Response Rate | Baseline until 60 days after last administration of CP-506
  Objective response rate (ORR) by RECIST 1.1 - the proportion of patients with a confirmed reduction in tumour burden of a predefined amount (this will include short lived responses).
Percentage change in tumour size | Baseline until 60 days after last administration of CP-506
  Percentage change in tumour size will be determined for patients with measurable disease at baseline and is derived at each visit by the percentage change from baseline in the sum of the diameters of target lesions. The best percentage change in tumour size will be the patient's value representing the largest decrease (or smallest increase) from baseline in tumour size

CONTACTS AND LOCATIONS:
Overall Officials: Loes Jansen, MD, Principal Investigator — Maastricht University Medical Center; Henk Verheul, MD, PhD, Principal Investigator — Erasmus Medical Center; Nuria Kotecki, MD, PhD, Principal Investigator — Jules Bordet Institute; Sylvie Rottey, MD, PhD, Principal Investigator — UZ Gent; Irene Brana, MD, PhD, Principal Investigator — Institut Vall d'Hebron
Locations (5):
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - UZ Gent, Ghent
- Netherlands (2):
  - Academisch Ziekenhuis Maastricht (Leading Centre), Maastricht, Limburg
  - Erasmus MC, Rotterdam
- Institut Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fu Z, Mowday AM, Smaill JB, Hermans IF, Patterson AV. Tumour Hypoxia-Mediated Immunosuppression: Mechanisms and Therapeutic Approaches to Improve Cancer Immunotherapy. Cells. 2021 Apr 24;10(5):1006. doi: 10.3390/cells10051006. PMID 33923305
- [Background] van der Wiel AMA, Jackson-Patel V, Niemans R, Yaromina A, Liu E, Marcus D, Mowday AM, Lieuwes NG, Biemans R, Lin X, Fu Z, Kumara S, Jochems A, Ashoorzadeh A, Anderson RF, Hicks KO, Bull MR, Abbattista MR, Guise CP, Deschoemaeker S, Thiolloy S, Heyerick A, Solivio MJ, Balbo S, Smaill JB, Theys J, Dubois LJ, Patterson AV, Lambin P. Selectively Targeting Tumor Hypoxia With the Hypoxia-Activated Prodrug CP-506. Mol Cancer Ther. 2021 Dec;20(12):2372-2383. doi: 10.1158/1535-7163.MCT-21-0406. Epub 2021 Oct 8. PMID 34625504
- [Background] Solivio MJ, Stornetta A, Gilissen J, Villalta PW, Deschoemaeker S, Heyerick A, Dubois L, Balbo S. In Vivo Identification of Adducts from the New Hypoxia-Activated Prodrug CP-506 Using DNA Adductomics. Chem Res Toxicol. 2022 Feb 21;35(2):275-282. doi: 10.1021/acs.chemrestox.1c00329. Epub 2022 Jan 20. PMID 35050609
- [Background] Jackson-Patel V, Liu E, Bull MR, Ashoorzadeh A, Bogle G, Wolfram A, Hicks KO, Smaill JB, Patterson AV. Tissue Pharmacokinetic Properties and Bystander Potential of Hypoxia-Activated Prodrug CP-506 by Agent-Based Modelling. Front Pharmacol. 2022 Feb 8;13:803602. doi: 10.3389/fphar.2022.803602. eCollection 2022. PMID 35211015
- [Derived] Yaromina A, Koi L, Schuitmaker L, van der Wiel AMA, Dubois LJ, Krause M, Lambin P. Overcoming radioresistance with the hypoxia-activated prodrug CP-506: A pre-clinical study of local tumour control probability. Radiother Oncol. 2023 Sep;186:109738. doi: 10.1016/j.radonc.2023.109738. Epub 2023 Jun 12. PMID 37315579
- See also: Holder of CP-506 IP — https://www.convertpharma.com/
- See also: Video of mechanism of action — https://youtu.be/1sidMh5ZF70